CLINICAL TRIAL: NCT02115945
Title: COMPARISON OF CONTINUOUS FEMORAL NERVE BLOCK AND PATIENT CONTROLLED EPIDURAL ANALGESIA AFTER TOTAL KNEE ARTHROPLASTY
Brief Title: Femoral and Epidural Block After Total Knee Arthroplasty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, MD, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SARI-01
Record Dates: First submitted 2014-04-08; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Acute Postoperative Pain; Chronic Postoperative Pain
Keywords: chronic postoperative pain; total knee arthroplasty; femoral block; We aimed to compare the effects of epidural and femoral block on acute and chronic postoperative pain.
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- epidural block (Experimental): Visual anlogue score vas used to evaluate pain. The anxiety/depression scale (HAD) was used to assess anxiety and depression. The SF 12 test (SHORT FORM 12) was used to evaluate quality of life. The DN4 test was used to evaluate neuropathic pain.
  Interventions: Other: DN4 test; Other: The SF 12 test; Other: HAD scale; Other: Visual analogue score; Procedure: epidural block
- femoral block (Active Comparator): Visual anlogue score vas used to evaluate pain. The anxiety/depression scale (HAD) was used to assess anxiety and depression. The SF 12 test (SHORT FORM 12) was used to evaluate quality of life. The DN4 test was used to evaluate neuropathic pain.
  Interventions: Other: DN4 test; Other: The SF 12 test; Other: HAD scale; Other: Visual analogue score; Procedure: femoral block

INTERVENTIONS:
Other: DN4 test — The DN4 test was used to evaluate neuropathic pain.
Other: The SF 12 test — The SF 12 test (SHORT FORM 12) was used to evaluate quality of life.
  Other Names: SHORT FORM 12
Other: HAD scale — The anxiety/depression scale (HAD) was used to assess anxiety and depression.
  Other Names: The anxiety/depression scale
Other: Visual analogue score — Visual analogue score vas used to evaluate pain.
  Other Names: VAS score
Procedure: femoral block
  Arms: femoral block
Procedure: epidural block
  Arms: epidural block

SUMMARY:
Total knee prosthetic replacement causes severe postoperative pain. Various analgesic techniques have been used in pain control. Comparison of epidural and femoral nerve block is lacking, furthermore effect on chronic pain is unclear. The investigators aimed to compare the effects of epidural and femoral block on acute and chronic postoperative pain.

DETAILED DESCRIPTION:
Background and aim Total knee prosthetic replacement causes severe postoperative pain. Various analgesic techniques have been used in pain control. Comparison of epidural and femoral nerve block is lacking, furthermore effect on chronic pain is unclear. The investigators aimed to compare the effects of epidural and femoral block on acute and chronic postoperative pain.

Methods The study was of randomized, prospective, and double-blind design and was conducted with 80 patients who had undergone total knee prosthetic replacement surgery with the insertion of a femoral nerve block or epidural block catheter to initiate postoperative analgesia. One-sided spinal anesthesia was performed in all the patients. Postoperative pain control was achieved with the administration via catheter using bupivacaine for patient-controlled analgesia. Acute postoperative pain was evaluated in the first 24 hours and chronic postoperative pain in the 1st and 3rd months following surgery. The anxiety/depression scale was used to assess anxiety and depression, the SF 12 test was used to evaluate quality of life, and the DN4 test was employed at patient visits at the 1st and 3rd months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of total knee arthroplasty

Exclusion Criteria:

* Patients with pain syndromes
* Patients using routinely medications for pain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Persistent surgical pain after total knee arthroplasty assessed by VAS scale | 3 months

SECONDARY OUTCOMES:
The anxiety and depression was evaluated with Hospital anxiety and depression scale. | 3 months

OTHER OUTCOMES:
Quality of life was evaluated with SF 12 test. | 3 months
Neuropathic pain was evaluated with DN4 test. | 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Sari, Assistant Prof, Study Chair — Adnan Menderes University Medical Faculty Anesthesiology and Reanimation Department; Fatma Şengül, MD, Principal Investigator — Antalya Education and Research Hospital, Anesthesiology and Reanimation Department, Antalya; Turkey; FabrizioGalimberti Galimberti, Medical Student, Principal Investigator — Cleveland ClinicLernerCollege of Medicine, Cleveland, Ohio; Bilge Karslı, Prof, Principal Investigator — Antalya Education and Research Hospital, Anesthesiology and Reanimation Department, Antalya; Turkey; Alparslan Turan, Associate Prof, Principal Investigator — Department of Outcomes Research, Cleveland Clinic; Murat Bakıs, Assistant Prof, Principal Investigator — Adnan Menderes University Medical Faculty, Anesthesiology and Reanimation Department, Aydin; Turkey
Locations (1):
- Adnan Menderes University Medical Faculty, Anesthesiology and Reanimation Department, Aydin, Turkey (Türkiye)

REFERENCES:
- [Result] Chan EY, Fransen M, Sathappan S, Chua NH, Chan YH, Chua N. Comparing the analgesia effects of single-injection and continuous femoral nerve blocks with patient controlled analgesia after total knee arthroplasty. J Arthroplasty. 2013 Apr;28(4):608-13. doi: 10.1016/j.arth.2012.06.039. Epub 2012 Nov 8. PMID 23142441